CLINICAL TRIAL: NCT00089635
Title: A Phase 2 Multicenter Single Arm Clinical Trial of ABX-EGF Monotherapy in Subjects With Metastatic Colorectal Cancer Whose Tumors Express Low or Negative EGFr Levels of Immunohistochemistry Following Treatment With Fluoropyrimidine, Irinotecan, and Oxaliplatin Chemotherapy
Brief Title: Panitumumab (ABX-EGF) Monotherapy in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030250; NCT00112944 (obsolete NCT alias)
Record Dates: First submitted 2004-08-09; First posted 2004-08-11 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer; Metastases
Keywords: Colon, Rectal Cancer; ABX-EGF, Panitumumab, EGFr; Immunex, Abgenix, Amgen; Metastatic Colorectal Cancer; Vectibix
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms | interventions — Panitumumab

ARMS (1):
- Panitumumab (Experimental): Panitumumab was administered by intravenous (IV) infusion at a dose of 6 mg/kg once every 2 weeks until participants developed progressive disease, were unable to tolerate investigational product, or discontinued for other reasons.
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — Administered by intravenous infusion
  Other Names: ABX-EGF; Vectibix®

SUMMARY:
The purpose of this study is to determine that panitumumab will have clinically meaningful anti-tumor activity in patients with metastatic colorectal cancer who have developed progressive disease or relapsed while on or after prior fluoropyrimidine, irinotecan and oxaliplatin chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of colorectal adenocarcinoma (diagnostic tissue obtained by tissue biopsy)
* Metastatic colorectal carcinoma
* Eastern Cooperative Oncology Group of 0, 1 or 2
* Documented evidence of disease progression during, or following treatment, with fluoropyrimidine, irinotecan and oxaliplatin chemotherapy for metastatic colorectal cancer
* Radiographic documentation of disease progression during or within 6 months following the most recent chemotherapy regimen is required
* Bidimensionally measurable disease
* Tumor expressing low to negative levels of epidermal growth factor receptor (EGFr) by immunohistochemistry
* At least 2 but no more than 3 prior chemotherapy regimens for metastatic colorectal cancer
* Adequate hematologic, renal and hepatic function

Exclusion Criteria:

* Symptomatic brain metastases requiring treatment
* Patient with a history of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis
* Use of systemic chemotherapy or radiotherapy within 30 days before enrollment
* Prior anti-EGFr antibody therapy with the exception of the small molecule EGFr tyrosine kinase inhibitors, which are permitted
* Prior anti-tumor therapies including prior experimental agents or approved anti-tumor small molecules and biologics of short (less than 1 week) serum half-life within 30 days before enrollment, or prior experimental or approved proteins within 6 weeks before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2004-08-01 (Actual); Primary Completion 2007-01-01 (Actual); Study Completion 2008-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Liao MZ, Prenen H, Dutta S, Upreti VV. The impact of hepatic and renal function on panitumumab exposures in patients with metastatic RAS wild-type colorectal cancer. Cancer Chemother Pharmacol. 2021 Oct;88(4):665-672. doi: 10.1007/s00280-021-04319-w. Epub 2021 Jul 2. PMID 34213592
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: FDA-approved Drug Labeling — http://www.vectibix.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 11 August 2004 through 2 August 2006
Period: Overall Study
Arm/Group | Panitumumab
Started | 203
Completed | 160
Not Completed | 43
Not completed — Adverse Event | 2
Not completed — Death | 17
Not completed — Disease Progression | 12
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 6
Not completed — Ineligibility determined | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Panitumumab
Number analyzed (Participants) | 203
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [54 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 114
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2
  Asian | 3
  Black or African American | 34
  Hispanic or Latino | 13
  White or Caucasian | 151

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Through Week 16
Description: Confirmed objective tumor response was defined as a complete response or partial response from enrollment through Week 16. Tumor response was monitored, beginning at Week 8, per a modified version of the World Health Organization (WHO) criteria for tumor response and progression by an independent review committee central assessment. Complete response was defined per modified WHO criteria as disappearance of all lesions (index and non-index). Partial response was defined as ≥ 50% decrease from Baseline in the sum of the products of the longest diameters (SPD) of index lesions. Scans were required to confirm a complete or partial response no earlier than 4 weeks from the time a response of complete or partial response was first documented.
Time Frame: From enrollment through Week 16
Population: Adjudicated Prior Failures Analysis Set, composed of all consented and enrolled participants who were determined to be eligible by the Independent Eligibility Review Committee (IERC).
Measure: Number; unit: participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 158
participants | 6

2. Primary Outcome: Duration of Response
Description: Kaplan-Meier estimate of time time from first objective response to first observed progression of disease or death if the death was due to disease progression (whichever comes first) among participants who had a response at any time on study. Participants who responded and did not progress while on study or who died for reasons other than disease progression while on study were censored at their last evaluable assessment date.
Time Frame: From enrollment until the data cut-off date of 22 December 2006. The median follow-up time was 36 weeks.
Population: Subset of Adjudicated Prior Failures Analysis Set, composed of all consented and enrolled participants who were determined to be eligible by the Independent Eligibility Review Committee (IERC), who had a confirmed objective tumor response at any time on study.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 7
weeks | 22.2 [16.1 to 28.4]

3. Secondary Outcome: Objective Tumor Response Throughout the Study
Description: Confirmed objective tumor response was defined as a complete response or partial response from enrollment through to the data cut-ff date. Tumor response was monitored, beginning at Week 8, per a modified version of the World Health Organization (WHO) criteria for tumor response and progression by an independent review committee central assessment. Complete response was defined per modified WHO criteria as disappearance of all lesions (index and non-index). Partial response was defined as ≥ 50% decrease from Baseline in the sum of the products of the longest diameters (SPD) of index lesions. Scans were required to confirm a complete or partial response no earlier than 4 weeks from the time a response of complete or partial response was first documented.
Time Frame: From enrollment until the data cut-off date of 22 December 2006. The median follow-up time was 36 weeks.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 158
participants | 7

4. Secondary Outcome: Time to Initial Objective Response
Description: Time from date of enrollment to first objective response; participants with stable disease at their last evaluable assessment date were censored at this date and participants with progressive disease while on study were censored after the last response was observed for all participants.
Time Frame: From enrollment until the data cut-off date of 22 December 2006. The median follow-up time was 36 weeks.
Population: Subset of Adjudicated Prior Failures Analysis Set, composed of all consented and enrolled participants who were determined to be eligible by the Independent Eligibility Review Committee (IERC), who had an objective tumor response at any time on study.
Measure: Median (Full Range); unit: weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 7
weeks | 11 [7 to 23]

5. Secondary Outcome: Progression-free Survival Time
Description: Kaplan-Meier estimate of median time from date of enrollment to date of first observed progression or death (whichever comes first); participants who did not progress while on study and did not die while on study were censored at their last evaluable assessment date.
Time Frame: From enrollment until the data cut-off date of 22 December 2006. The median follow-up time was 36 weeks.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 158
weeks | 8.1 [7.4 to 11.3]

6. Secondary Outcome: Time to Disease Progression
Description: Kaplan-Meier estimate of median time from date of enrollment to date of first observed progression or death date if the death was due to disease progression (whichever comes first); participants who have not progressed while on study or died for reasons other than disease progression while on study were censored at their last evaluable assessment date.
Time Frame: From enrollment until the data cut-off date of 22 December 2006. The median follow-up time was 36 weeks.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 158
weeks | 8.3 [7.4 to 11.3]

7. Secondary Outcome: Time to Treatment Failure
Description: Kaplan-Meier estimate of median time from date of enrollment to date decision was made to end the treatment phase for any reason; participants who complete the treatment phase or who remain in the treatment phase at the completion of the study were censored at this time.
Time Frame: From enrollment until the data cut-off date of 22 December 2006. The median follow-up time was 36 weeks.
Population: Subset of Adjudicated Prior Failures Analysis Set, composed of all consented and enrolled participants who were determined to be eligible by the Independent Eligibility Review Committee (IERC), for whom a decision was made to end treatment for any reason.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 158
weeks | 8.4 [8.1 to 11.3]

8. Secondary Outcome: Duration of Stable Disease
Description: Kaplan-Meier estimate of median time from date of enrollment to date of first observed progression or death date if the death was due to disease progression (whichever comes first); in those participants who had a best response of stable disease.
  Stable Disease is defined as neither sufficient shrinkage of index lesions to qualify for a partial response nor sufficient increase to qualify for progressive disease taking as reference the nadir sum of the products of the longest diameters since the treatment started.
Time Frame: From enrollment until the data cut-off date of 22 December 2006. The median follow-up time was 36 weeks.
Population: Subset of Adjudicated Prior Failures Analysis Set, composed of all consented and enrolled participants who were determined to be eligible by the Independent Eligibility Review Committee (IERC), who had a best response of stable disease.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 52
weeks | 16.0 [15.3 to 22.9]

9. Secondary Outcome: Overall Survival
Description: Kaplan-Meier estimate of time to death from any cause; participants who had not died while on study or were lost to follow-up were censored at their last contact date.
Time Frame: From enrollment until the data cut-off date of 22 December 2006. The median follow-up time was 36 weeks.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 158
months | 9.0 [8.1 to 11.2]

ADVERSE EVENTS:
Time Frame: First dose date through the safety follow-up visit. The median time frame is 2.6 months.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Panitumumab
Serious Adverse Events (participants affected / at risk) | 61/203
Other Adverse Events (participants affected / at risk) | 200/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab (N=203)
Anaemia (Blood and lymphatic system disorders) | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Pancreatitis (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Infusion related reaction (General disorders) | 2
Pyrexia (General disorders) | 4
Bile duct obstruction (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Anaphylactic reaction (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Klebsiella bacteraemia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Prothrombin time prolonged (Investigations) | 1
Urine output decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Failure to thrive (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab (N=203)
ANAEMIA (Blood and lymphatic system disorders) | 14
CONJUNCTIVITIS (Eye disorders) | 11
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 13
ABDOMINAL PAIN (Gastrointestinal disorders) | 31
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 14
CONSTIPATION (Gastrointestinal disorders) | 34
DIARRHOEA (Gastrointestinal disorders) | 55
NAUSEA (Gastrointestinal disorders) | 68
STOMATITIS (Gastrointestinal disorders) | 15
VOMITING (Gastrointestinal disorders) | 53
ASTHENIA (General disorders) | 19
FATIGUE (General disorders) | 71
OEDEMA PERIPHERAL (General disorders) | 26
PYREXIA (General disorders) | 19
PARONYCHIA (Infections and infestations) | 42
RASH PUSTULAR (Infections and infestations) | 18
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11
WEIGHT DECREASED (Investigations) | 24
ANOREXIA (Metabolism and nutrition disorders) | 44
DEHYDRATION (Metabolism and nutrition disorders) | 13
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 11
HYPOKALAEMIA (Metabolism and nutrition disorders) | 14
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 28
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15
BACK PAIN (Musculoskeletal and connective tissue disorders) | 21
DIZZINESS (Nervous system disorders) | 14
HEADACHE (Nervous system disorders) | 18
NEUROPATHY PERIPHERAL (Nervous system disorders) | 11
ANXIETY (Psychiatric disorders) | 14
DEPRESSION (Psychiatric disorders) | 11
INSOMNIA (Psychiatric disorders) | 19
COUGH (Respiratory, thoracic and mediastinal disorders) | 28
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 33
ACNE (Skin and subcutaneous tissue disorders) | 11
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 141
DRY SKIN (Skin and subcutaneous tissue disorders) | 41
ERYTHEMA (Skin and subcutaneous tissue disorders) | 137
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 48
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 12
PRURITUS (Skin and subcutaneous tissue disorders) | 140
RASH (Skin and subcutaneous tissue disorders) | 59
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 14
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 23
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.